CLINICAL TRIAL: NCT01488812
Title: Waiting Time to Operation for Hip-fracture Patients
Status: Completed | Type: Observational
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Olof Skoldenberg, Consultant Orthopaedic Surgeon, Danderyd Hospital
Other Study IDs: 2010/2029-32
Record Dates: First submitted 2011-12-07; First posted 2011-12-08 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Hip-fracture
Keywords: Hip-fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hip-fracture patients: All the hip-fracture patients admitted to the Orthopaedic Depart of Danderyd Hospital between 1st June 2007- 1st June 2008 who fulfilled the inclusion criteria of the study.

SUMMARY:
This study investigates the relationship between waiting time to surgery and the risk for medical complications and 1-year mortality in hip-fracture patients.

ELIGIBILITY:
Inclusion Criteria:

* Hip-fracture patient

Exclusion Criteria:

* Periprosthetic fracture
* Pathological fracture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hip fracture patients admitted to Danderyd Hospital Orthopaedic Department from 1st June 2007 to 1st June 2008
Sampling Method: Non-Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olof Skoldenberg, Principal Investigator — Danderyd Hospital, Stockholm, Sweden
Locations (1):
- Danderyd Hospital, Stockholm, Sweden